CLINICAL TRIAL: NCT03441529
Title: A Phase 1, Open-label, Randomized, 2-period, Crossover Study to Assess the Effect of Intravenous Infusion of Piperacillin/Tazobactam on the Pharmacokinetics of Orally Administered Lumicitabine (JNJ-64041575) in Healthy Adult Subjects
Brief Title: A Crossover Study to Assess the Effect of Intravenous Infusion of Piperacillin/Tazobactam on the Pharmacokinetics of Orally Administered Lumicitabine (JNJ-64041575) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108431; 2017-004504-22 (EudraCT Number); 64041575RSV1009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Healthy
MeSH Terms: interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1 (AB) (Experimental): Participants will receive Treatment A as a single oral dose of 1000 milligram (mg) lumicitabine (4*250 mg tablets) on Day 1 of period 1 followed by Treatment B as a single oral dose of 1000 mg lumicitabine (4*250 mg tablets) together with piperacillin/tazobactam administered as three 30-minute Intravenous (IV) infusions of 4.5 gram (g) piperacillin/tazobactam (4 g of piperacillin and 0.5 g of tazobactam) every 6 hours on Day 1 of period 2. A washout period of at least 21 days will be maintained between each treatment period.
  Interventions: Drug: Lumicitabine; Drug: Piperacillin/Tazobactam
- Treatment Sequence 2 (BA) (Experimental): Participants will receive Treatment B on Day 1 of period 1 followed by Treatment A on Day 1 of period 2. A washout period of at least 21 days will be maintained between each treatment period.
  Interventions: Drug: Lumicitabine; Drug: Piperacillin/Tazobactam

INTERVENTIONS:
Drug: Lumicitabine — Participants will receive single oral dose of 1000 mg lumicitabine as per assigned treatment sequence.
  Other Names: JNJ-64041575, ALS-008176
Drug: Piperacillin/Tazobactam — Participants will receive three IV infusions of piperacillin/tazobactam combination product (4 g of piperacillin and 0.5 g of tazobactam) every 6 hours on Day 1.

SUMMARY:
The main purpose of this study is to evaluate the effect of intravenous (IV) infusions of piperacillin/tazobactam on the pharmacokinetics (PK) of JNJ-63549109 after a single oral dose of lumicitabine in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI); weight in kg divided by the square of height in meters) between 18.0 and 30.0 kilogram per square meter (kg/m^2), extremes included, and a body weight not less than 50.0 kg, inclusive, at screening
* Participant must have a blood pressure between 90 and 140 millimeter of mercury (mmHg) systolic, extremes included, and no higher than 90 mmHg diastolic. If blood pressure is out of range, 1 repeated assessment is permitted after an additional 5 minutes of rest
* Participants must have normal values for alanine transaminase (ALT) and aspartate aminotransferase (AST) (less than or equal to [<=] 1.0*upper limit of laboratory normal range [ULN])
* Participant must have a normal renal function (estimated glomerular filtration rate [eGFR] greater than or equal to [>=] 90 milliliter per minute per 1.73 square meter [mL/min/1.73m^2]) determined by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
* A female Participant, except if postmenopausal, must have a negative serum beta human chorionic gonadotropin (beta hCG) pregnancy test at screening, and a negative urine beta hCG pregnancy test on Day 1 of each treatment period
* Participant must be healthy on the basis of medical history, physical examination, 12 lead electrocardiogram (ECG), vital signs, and laboratory tests performed at screening

Exclusion Criteria:

* Participant has a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease (example, glucose 6 phosphate dehydrogenase deficiency), coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, seizure disorders, or any other illness, that in the investigator's and/or sponsor's medical monitor opinion should exclude the participant or that could interfere with the interpretation of the study results
* Participant has a history of human immunodeficiency virus type 1 (HIV-1) or type 2 (HIV-2) antibody positive, or tests positive for HIV-1 or -2 at screening
* Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well being) or that could prevent, limit, or confound the protocol specified assessments
* Participants with a history of allergic reactions to any of the penicillins, cephalosporins, monobactams, carbapenems, or beta lactamase inhibitors (clavulanate, sulbactam, tazobactam, avibactam), or other contra indications for the use of piperacillin/tazobactam
* Participant with a history of clinically significant drug allergy such as, but not limited to, sulfonamides, or drug allergy diagnosed in previous studies with experimental drugs
* Participant has known allergies, hypersensitivity, or intolerance to lumicitabine or its excipients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-63549109 (Metabolite of JNJ-64041575) | Predose, 15 minutes (min), 30 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  Cmax is the maximum observed plasma concentration.
Area Under Plasma Concentration Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of JNJ-63549109 (Metabolite of JNJ-64041575) | Predose, 15 min, 30 min, 1h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  Area under the plasma concentration time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-63549109 (Metabolite of JNJ-64041575) | Predose, 15 min, 30 min, 1h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/ lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-63549109 (Metabolite of JNJ- 64041575) | Predose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  Tmax is the actual sampling time to reach maximum observed plasma concentration.
Observed Plasma Concentration at 12 Hours Post dose (C12h) of JNJ-63549109 (Metabolite of JNJ- 64041575) | 12 hours postdose
  C12h is observed plasma concentration at 12 hours post dose.
Observed Plasma Concentration at 24 Hours Post dose (C24h) of JNJ-63549109 (Metabolite of JNJ- 64041575) | 24 hours postdose
  C24h is observed plasma concentration at 24 hours post dose.
Elimination Rate Constant (Lambda[z]) of JNJ-63549109 (Metabolite of JNJ- 64041575) | Predose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  Lambda[z] is the apparent terminal elimination rate constant, estimated by linear regression using the terminal logarithmic (log)-linear phase of the log-transformed concentration vs time data.
Elimination Half-Life (T1/2) of JNJ-63549109 (Metabolite of JNJ- 64041575) | Predose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  T1/2 is the apparent terminal elimination half-life, calculated as 0.693/Lambda(z).

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-64167896 (Metabolite of JNJ-64041575) | Predose, 15 min, 30 min, 1h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  Cmax is the maximum observed plasma concentration.
Area Under Plasma Concentration Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of JNJ-64167896 (Metabolite of JNJ-64041575) | Predose, 15 min, 30 min, 1h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  Area under the plasma concentration time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-64167896 (Metabolite of JNJ-64041575) | Predose, 15 min, 30 min, 1h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/ lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to end of study (approximately 2 months)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ 64167896 (Metabolite of JNJ-64041575) | Predose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  Tmax is the actual sampling time to reach maximum observed plasma concentration.
Observed Plasma Concentration at 12 Hours Post dose (C12h) of JNJ 64167896 (Metabolite of JNJ-64041575) | 12 hours postdose
  C12h is observed plasma concentration at 12 hours post dose.
Observed Plasma Concentration at 24 Hours Post dose (C24h) of JNJ 64167896 (Metabolite of JNJ-64041575) | 24 hours postdose
  C24h is observed plasma concentration at 24 hours post dose.
Elimination Rate Constant (Lambda[z]) of JNJ 64167896 (Metabolite of JNJ-64041575) | Predose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  Lambda[z] is the apparent terminal elimination rate constant, estimated by linear regression using the terminal logarithmic (log)-linear phase of the log-transformed concentration vs time data.
Elimination Half-Life (T1/2) of JNJ 64167896 (Metabolite of JNJ-64041575) | Predose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 hours and end of study (16 days after last study drug intake or early withdrawal) (approximately 2 months)
  T1/2 is the apparent terminal elimination half-life, calculated as 0.693/Lambda(z).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium